CLINICAL TRIAL: NCT00061880
Title: Phase 1-2 Multi-Center Study of Intravenous BCX-1777 in Patients With Refractory Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: BCX-1777 in Treating Patients With Refractory Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: BIOCRYST-1777BC-103; CDR0000301763 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2004-07

CONDITIONS: Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

INTERVENTIONS:
Drug: forodesine hydrochloride

SUMMARY:
RATIONALE: BCX-1777 may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase I/II trial to study the effectiveness BCX-1777 in treating patients who have refractory cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of BCX-1777 in patients with refractory cutaneous T-cell lymphoma.
* Determine the efficacy of this drug in these patients.
* Determine the toxicity profile of this drug in these patients.
* Correlate plasma concentration of deoxyguanosine with clinical response and toxicity in patients treated with this drug.
* Determine the provisional optimal biological dose of this drug in these patients.

OUTLINE: This is an open-label, nonrandomized, dose-escalation, multicenter study.

* Phase I: Patients receive BCX-1777 IV over 30 minutes every 12 hours on days 1-5 (a total of 9 doses). Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BCX-1777 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive treatment as in phase I at the MTD of BCX-1777. Patients (including those who respond to treatment) are followed at 14 and 30 days, monthly for 6 months, every 2 months for 6 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 3-64 patients (3-24 for phase I and 40 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma (CTCL)

  * Any stage except IA patch only
* Previously treated according to 1 of the following:

  * Stage IA plaque, IB, or IIA:

    * At least 4 prior conventional and/or experimental regimens (topical or systemic, including psoralen-ultraviolet light [PUVA] and systemic corticosteroids)
  * Stage IIB, III, or IV:

    * At least 1 prior systemic regimen (systemic corticosteroids and PUVA do not count as systemic regimens for this purpose) NOTE: Repeated use of the same regimen is considered one regimen
* Measurable disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count at least 2,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (unless due to Gilbert's syndrome)
* ALT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* No hepatitis B or C

Renal

* Creatinine clearance at least 45 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Human T-cell leukemia virus type 1 (HTLV-1) negative
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other illness that would limit study participation
* No active serious infection not controlled by antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent anticancer antibody therapy
* No concurrent anticancer immunotherapy
* No concurrent anticancer gene therapy
* No concurrent anticancer vaccine therapy
* No concurrent anticancer angiogenesis inhibitors
* No concurrent sargramostim (GM-CSF)
* No concurrent filgrastim (G-CSF) during course 1 of therapy

Chemotherapy

* More than 21 days since prior chemotherapy unless fully recovered
* No concurrent anticancer chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 2 weeks since prior topical corticosteroids
* No concurrent anticancer hormonal therapy

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 2 weeks since prior antineoplastic therapy
* More than 21 days since prior investigational agents unless fully recovered
* No concurrent citrate-blood products within 30 minutes before or after study treatment
* No concurrent anticancer matrix metalloprotease inhibitors
* No other concurrent anti-CTCL therapy
* No concurrent use of tanning beds
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Shalaurov, MD, PhD, Study Chair — Inveresk Research Group, Incorporated
Locations (3):
- United States (3):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - University of Texas - MD Anderson Cancer Center, Houston, Texas